CLINICAL TRIAL: NCT06152601
Title: Early Standing in Children and Adolescent Operated on for Idiopathic Scoliosis
Brief Title: Early Standing in Minors Operated on for Idiopathic Scoliosis
Acronym: LevPOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/21/0611
Record Dates: First submitted 2023-09-13; First posted 2023-11-30 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Idiopathic Scoliosis; ERAS
Keywords: idiopathic scoliosis; physiotherapies; ERAS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group experimental (Experimental): Patient between 12 and 18 years old with a spinal surgery for idiopathic scoliosis programmed. Immediately postoperatively, during his stay in a PACU or ICU, the patient will be offered a physiotherapy session including a lifting phase in a bipedal standing position.
  Interventions: Procedure: anticipated bipedal standing position in the immediate post-operative phase

INTERVENTIONS:
Procedure: anticipated bipedal standing position in the immediate post-operative phase — Realization of a first stand-up within 6 hours after entry into PACU or extubation for admitted patients intubated, in PACU or on admission to ICU by a state-certified physiotherapist.
  Immediately postoperatively, during his stay in a Intensive Care Unit, the patient will be offered a physiotherapy session including a lifting phase in a bipedal standing position.

SUMMARY:
The implementation of an enhanced rehabilitation after surgery (ERAS) program in major orthopedic surgery and in scoliosis surgery in children and adolescents has become a marker of good practice. Investigators are already applying anesthetic, surgical, peri-operative medicine and rehabilitation techniques allowing accelerated and improved rehabilitation for scoliosis operated patients in the establishment. To improve patient care, the Investigators want to develop the ERAS program. The objective of this research will be to validate the feasibility of getting up early on D0 in post-anesthesia care unit (PACU) or ICU in children who have just had surgery for idiopathic scoliosis.

DETAILED DESCRIPTION:
The study hypothesize that entry into an early mobilizing physiotherapy program, i.e., from the immediate postoperative period, from the PACU or the ICU, could improve the outcome of patients in terms of pain, anxiety, re-empowerment, length of stay and ultimately overall satisfaction.

Following a general anesthesia, the patient is monitored in the PACU the time to recover respiratory, neurological and hemodynamic autonomy. It is also in PACU that the team optimize pain management, through opioid treatments if necessary.

The first physiotherapy sessions including sitting on the edge of the bed and getting up for the first time are technical acts that require good cooperation from the patient and adequate pain relief. Usually, physiotherapy rehabilitation is started on the first postoperative day. However, once the stability of vital functions and the analgesia have been optimized, the early postoperative phase seems to be a privileged moment to begin this rehabilitation program. This early physiotherapy treatment could also have a beneficial psychological effect on the rest of the treatment.

Although most centers tend to generalize ERAS programs and early rehabilitation techniques, to date there is no publication on the feasibility of early rehabilitation from the immediate postoperative period, nor on the expected benefit of such a program. The fact of starting the rehabilitation immediately postoperatively or as soon as the PACU could have several advantages. The optimization of pain management performed in the PACU could facilitate the physiotherapy session. In addition, it turns out that the rehabilitation and progressive re-empowerment of the patient have a positive psychological and physical effect on the rest of the treatment. The early re-empowerment of the patient allows him to regain control of his body and his care which has a positive psychological effect on the care. Early mobilization fights muscle contracture with positive effects on pain and patient comfort.

This research propose to validate the feasibility of standing up early on D0 in PACU or ICU in children who have just had surgery for idiopathic scoliosis. Immediately postoperatively, during his stay in a PACU or ICU, the patient will be offered a physiotherapy session including a lifting phase in a bipedal standing position.

ELIGIBILITY:
Inclusion Criteria:

* Programming of spinal surgery via the posterior approach for idiopathic scoliosis eligible for an ERAS program
* Person affiliated or beneficiary of a social security scheme
* Free, informed and written consent signed by the legal guardians of the minor patient
* Free and informed consent of the minor patient

Exclusion Criteria:

* Scoliosis linked to a neuromuscular pathology
* Physical status score of American Society of Anesthesiologists (ASA) > 2
* Severe or unbalanced associated conditions (cardiac, pulmonary, coagulopathy or anticoagulant treatment with curative intent, long-term corticosteroid therapy)
* Malnutrition
* Major cognitive disorders
* Impossibility for the parent(s) to contact the pediatrician or the hospital service if necessary (minor patients)
* Pregnancy
* Feeding with milk
* Severe disability related to scoliosis with impossibility of ambulation
* Surgical assembly planned unstable or requiring the wearing of a corset
* Refusal of minor patient or of the legal guardians of the minor patient
* Patient under legal protection, guardianship or curatorship

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
success of the anticipated bipedal standing position within 6 hours postoperative | Hour 6
  success of a Stand up in a bipedal standing position during more than 3 seconds in the post-operative phase within 6 hours postoperative. The procedure of anticipated bipedal standing position is realised according to the same procedure as usual but carried out in advance, at six hours postoperative, after validation of the prerequisites for the procedure.

SECONDARY OUTCOMES:
pain measured by visual analog scale at baseline | day 0
  pain measured by visual analog scale at baseline. The visual analog scale measure the pain from 0 to 10. 0 means no pain and 10 means the worst possible pain
pain measured by visual analog scale at the first day postoperative | day 1
  pain measured by visual analog scale at the first day postoperative. The visual analog scale measure the pain from 0 to 10. 0 means no pain and 10 means the worst possible pain
pain measured by visual analog scale at the second day postoperative | day 2
  pain measured by visual analog scale at the second day postoperative. The visual analog scale measure the pain from 0 to 10. 0 means no pain and 10 means the worst possible pain
pain measured by visual analog scale at the third day postoperative | day 3
  pain measured by visual analog scale at the third day postoperative. The visual analog scale measure the pain from 0 to 10. 0 means no pain and 10 means the worst possible pain
Morphine consumption baseline | Day 0
  consumption in morphine per day
Morphine consumption at Day 1 | Day 1
  consumption in morphine per day
Morphine consumption at Day 2 | Day 2
  consumption in morphine per day
Morphine consumption at Day 3 | Day 3
  consumption in morphine per day
Postoperative length of stay | Day 7
  Postoperative length of stay
success of the anticipated bipedal standing position in the early post operative phase (within 2 hours postoperative) | Hour 2
  success of a Stand up in a bipedal standing position during more than 3 seconds in the immediate post-operative phase (i.e., within 2 hours postoperative). The procedure of anticipated bipedal standing position is realised according to the same procedure as usual but carried out in advance, in the early post operative phase in the post-anesthesia care unit (PACU), after validation of the prerequisites for the procedure.
success of the anticipated bipedal standing position in the early post operative phase (within 3 hours postoperative) | Hour 3
  success of a Stand up in a bipedal standing position during more than 3 seconds in the post-operative phase (i.e., within 3 hours postoperative). The procedure of anticipated bipedal standing position is realised according to the same procedure as usual but carried out in advance, in the early post operative phase in the post-anesthesia care unit (PACU), after validation of the prerequisites for the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: François Dr DELORT, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de TOULOUSE, Toulouse, France